CLINICAL TRIAL: NCT01501123
Title: Re-hospital Agitation and Sedation Trial: A Randomized Controlled Trial of Haloperidol Versus Midazolam for the Sedation of the Agitated Patient
Brief Title: Pre-hospital Agitation and Sedation Trial: A Randomized Controlled Trial of Haloperidol Versus Midazolam for the Sedation of the Agitated Patient
Acronym: PHAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic Health East (Other)
Responsible Party: Principal Investigator, Derek Isenberg, MD, Catholic Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCMC 2010-24
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Agitation
Keywords: Time to sedation of agitated patients
MeSH Terms: conditions — Psychomotor Agitation | interventions — Haloperidol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haloperidol (Experimental): IM Haloperidol
  Interventions: Drug: Haloperidol
- IM Midazolam (Active Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Haloperidol — 5mg IM
  Arms: Haloperidol
Drug: Midazolam — IM midazolam
  Arms: IM Midazolam

SUMMARY:
PREHOSPITAL AGITATION AND SEDATION TRIAL (PHAST)

* The goal of the PHAST is to demine whether haloperidol is superior to midazolam for the sedation of agitated patients in the prehospital environment
* The primary outcome is the time to a Richmond Agitation and Sedation Scale (RASS) ≤1

  o The RASS is a well validated standardized score to measure a patient's agitation
* The secondary outcomes are

  * Time until RASS returns to 0 or 1 if RASS <0
  * Need for additional sedation
  * Adverse effects (need for intubation, arrhythmia)
* Mercy EMS will be the only EMS agency in the Commonwealth of Pennsylvania carrying haloperidol
* Identification of potential study patients will be per state protocols
* Exclusion Criteria for the study
* Age <18
* Pregnant
* Allergic to study medication
* Transport to hospital other than Mercy Fitzgerald Hospital
* Unable to reach medical command prior to giving medication
* When a paramedic identifies a possible study candidate, the paramedic will consult medical command to see if the patient is appropriate for the study
* If the medical command agrees the patient is appropriate for the study, patients will be randomized to
* Odd days: Haloperidol 5mg IM (age <65) or haloperidol 2.5 mg IM (age ≥65)
* Even days: Midazolam 0.05 mg IM to maximum of 5mg IM (age <65) or maximum of 2.5mg (age ≥65)
* The RASS will be documented by the prehospital providers every 5 minutes until arrival at the hospital
* Once the patient arrives at the ED, the RASS will be documented in PICIS® by the emergency department nurse at the time of triage and at a minimum of hourly until the RASS =0 or 1 for 2 consecutive hours
* Questions may be directed to Dr. Isenberg at disenberg@mercyhealth.org or at (267) 205-6453

Richmond Agitation Sedation Scale

RASS RASS Description

* 4 Combative, violent, danger to staff
* 3 Pulls or removes tube(s) or catheters; aggressive
* 2 Frequent non-purposeful movement
* 1 Anxious, apprehensive, but not aggressive 0 Alert and calm

  * 1 Awakens to voice (eye opening/contact) >10 sec
  * 2 Light sedation, briefly awakens to voice (eye opening/contact) <10 sec
  * 3 Moderate sedation, movement or eye opening. No eye contact
  * 4 Deep sedation, no response to voice, but movement or eye opening to physical stimulation
  * 5 Unarousable, no response to voice or physical stimulation

ELIGIBILITY:
Exclusion Criteria:

* Age <18
* Pregnant
* Allergic to study medication
* Transport to hospital other than Mercy Fitzgerald Hospital
* Unable to reach medical command prior to giving medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to sedation | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Derek Isenberg, MD, Principal Investigator — Mercy Catholic Medical Center
Locations (1):
- Mercy Catholic Medical Center, Darby, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No